CLINICAL TRIAL: NCT07070830
Title: Feasibility of Simplified Onboarding in Adults With Type 2 Diabetes Using Automated Insulin Delivery
Brief Title: Simplified Onboarding in Adults With Type 2 Diabetes
Acronym: SIMPLEUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIMPLEUSE
Record Dates: First submitted 2025-06-26; First posted 2025-07-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: T2D; Type 2 Diabetes; Omnipod; Omnipod 5; Automated Insulin Delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Omnipod M System with lower starting dose (Active Comparator)
  Interventions: Device: Active Comparator: Omnipod M System with lower starting dose
- Omnipod M System with higher starting dose (Active Comparator)
  Interventions: Device: Active Comparator: Omnipod M System with higher starting dose

INTERVENTIONS:
Device: Active Comparator: Omnipod M System with lower starting dose — Omnipod M Automated Insulin Delivery System with Dexcom G6 continuous glucose monitoring system
  Arms: Omnipod M System with lower starting dose
Device: Active Comparator: Omnipod M System with higher starting dose — Omnipod M Automated Insulin Delivery System with Dexcom G6 continuous glucose monitoring system
  Arms: Omnipod M System with higher starting dose

SUMMARY:
This is an outpatient study testing different starting doses of insulin in participants with type 2 diabetes. Participants will manage their diabetes using the Omnipod M System. The system is comprised of an Omnipod M Pod, an Omnipod M Controller, and will be used with a Dexcom G6 continuous glucose monitoring sensor (CGM). The main objectives of the study are to evaluate the safety and tolerability of different starting doses of insulin using the Omnipod M System.

There is a precursory evaluation before the main, randomized trial. Participation in the precursory evaluation could last up to 12 weeks and participation in the randomized trial could last up to 6 weeks. During both the evaluation and the randomized trial, participants will manage their diabetes using the Omnipod M System in Automated Mode.

An optional 12-weeks of continued Omnipod M System use is available upon completion of the randomized trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent 18-75 years
2. Diagnosed with type 2 diabetes, on current insulin regimen for at least 3 months prior to screening (i.e. Basal-bolus, basal only or pre-mix)
3. Basal-bolus (non-AID pump & MDI), pre-mix, or basal only users suitable for conversion to AID pump therapy for at least 3 months prior to screening. For basal-bolus and premix users, they must have A1c <14%. For basal only users must have A1c >7% and <14%.
4. Willing to use only the following types of U-100 insulin during the study: Humalog U-100, Novolog, Admelog, or their generic equivalents.
5. Participant agrees to provide their own insulin for the duration of the study
6. Stable doses over the preceding 4 weeks of other glucose-lowering medications as determined by Investigator
7. Stable doses of weight loss medications over the preceding 4 weeks, and plans to maintain throughout the study, that may affect glycemic control directly and/or indirectly, except for a dose reduction or discontinuation, as determined by Investigator
8. Willing to wear the system continuously throughout the study
9. Participant agrees to provide their own compatible smartphone for use with the Dexcom G6 CGM
10. Investigator has confidence that the participant has the cognitive ability and can successfully operate all study devices and can adhere to the protocol
11. Able to read and understand English
12. Willing and able to sign the Informed Consent Form (ICF)
13. If female of childbearing potential, willing and able to have pregnancy testing

Exclusion Criteria:

1. Use of an AID pump in automated mode up to 90 days prior to screening
2. Any medical condition which in the opinion of the Investigator, would put the participant at an unacceptable safety risk, such as untreated malignancy, unstable cardiac disease, unstable or end-stage renal disease, and/or eating disorders (i.e. anorexia/bulimia)
3. Arrhythmias or other cardiac conditions confirmed by ECG (within past 30 days) which in the opinion of the Investigator, would put the participant at an unacceptable safety risk
4. Current or known history of coronary artery disease that is not stable with medical management, including unstable angina, or angina that prevents moderate exercise despite medical management, or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting within the 12 months prior to screening
5. Any planned surgery during the study which could be considered major in the opinion of the Investigator
6. History of more than 1 severe hypoglycemic event in 6 months prior to screening
7. History of more than 1 episode of diabetic ketoacidosis (DKA) or hyperosmolar hyperglycemic syndrome (HHS) in the 6 months prior to screening; unrelated to an intercurrent illness; kinked, dislodged, or occluded cannula; or initial diabetes diagnosis
8. Blood disorder or dyscrasia within 3 months prior to screening, which in the Investigator's opinion could interfere with determination of HbA1c
9. Use of hydroxyurea
10. Has taken systemic steroids (oral or injectable) within 4 weeks or has had a local steroid injection (intraarticular, epidural) within 1 week prior to screening or plans to take oral or injectable steroids during the study
11. Unable to tolerate adhesive tape or has any unresolved skin condition that could impact sensor or pump placement
12. Pregnant or lactating, planning to become pregnant during the study, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable includes abstinence, condoms, oral/injectable contraceptives, IUD, or implant); childbearing potential means that menstruation has started, and the participant is not surgically sterile or greater than 12 months post-menopausal)
13. Planned international travel during the study
14. Participation in another clinical study using an investigational drug or device other than the Omnipod in the 30 days prior to screening or intends to participate during the study period
15. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the Investigator's clinical judgment
16. Participant is an employee of Insulet, an Investigator or Investigator's study team, or immediate family member (spouse, biological or legal guardian, child, sibling, parent) of any of the aforementioned

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Percent of time >180 mg/dL | Comparing baseline to days 7, 14, 21, and 28 and end of continuation phase in the randomized trial.
  Glucose metric from study continuous glucose monitoring system
Percent of time <70 mg/dL | Comparing baseline to days 7, 14, 21, and 28 and end of continuation phase in the randomized trial.
  Glucose metric from study continuous glucose monitoring system

SECONDARY OUTCOMES:
Percent of time in range (TIR) 70-180 mg/dL | Comparing baseline to days 7, 14, 21, and 28 and end of continuation phase in the randomized trial.
  Glucose metric from study continuous glucose monitoring system
Percent of time above range (TAR) >250 mg/dL | Comparing baseline to days 7, 14, 21, and 28 and end of continuation phase in the randomized trial.
  Glucose metric from study continuous glucose monitoring system
Percent of time below range (TBR) <54 mg/dL | Comparing baseline to days 7, 14, 21, and 28 and end of continuation phase in the randomized trial.
  Glucose metric from study continuous glucose monitoring system
Total daily insulin (TDI) | Comparing baseline to days 7, 14, 21, and 28 and end of continuation phase in the randomized trial.
  Glucose metric from study continuous glucose monitoring system
Total daily insulin/kg | Comparing baseline to days 7, 14, 21, and 28 and end of continuation phase in the randomized trial.
  Glucose metric from study continuous glucose monitoring system
Perception questionnaire | Comparing baseline to days 7, 14, 21, and 28 and end of continuation phase in the randomized trial.
  Includes questions about participant's private attitudes, feelings, and behavior related to the investigational device as well as managing diabetes.
Weight | Comparing baseline to end of continuation phase in the randomized trial.
  Measures change in weight
HbA1c | Comparing baseline to end of continuation phase in the randomized trial.
  Measures changes in HbA1c

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Colorado, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Joslin Diabetes Center, Boston, Massachusetts
  - MassResearch LLC., Waltham, Massachusetts
  - AccellaCare, Wilmington, North Carolina
  - Disease & Glandular Disease Clinic, San Antonio, Texas